CLINICAL TRIAL: NCT02373384
Title: The Predictors of Successful Oral Dissolution Therapy in Radiolucent Renal Stones; A Prospective Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Resident in Urology, Urology and Nephrology Center, Mansoura University, Mansoura, Egypt, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEl-Sawy122015
Record Dates: First submitted 2015-02-13; First posted 2015-02-27 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Urolithiasis; Renal Stones
Keywords: Radiolucent renal stones; Oral dissolution therapy; Systemic chemolysis; Renal uric acid stones; Alkalinization
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis | interventions — Potassium Citrate; Allopurinol; Red Meat; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group (Experimental): Eligible patients, who fulfilled the study criteria, will be instructed For;
  1. Oral alkalinization
     * Potassium citrate 20 mEq three times daily
     * Hyperuricosuric patients (24-hours urine uric acid more than 750 mg/day in male and more than 650mg/day in females), will receive Allopurinol, a competitive inhibitor of xanthine oxidase, in a dose of 300 mg daily.
  2. Life style modification Adequate fluid intake in order to maintain urine volume between 2-3 L per day.
  3. Dietary recommendations
  In hyperuricosuric patients (24-hours urine uric acid more than 750 mg/day in male and more than 650mg/day in females) ;
  - Dietary modification will be advised in the form of decrease purine rich diet as red meat and fish, increase vegetables.
  Interventions: Drug: Oral alkalinization (Potassium citrate, Allopurinol); Behavioral: Life style modification; Dietary Supplement: Dietary recommendations (decrease purine rich diet as red meat and fish, increase vegetables)

INTERVENTIONS:
Drug: Oral alkalinization (Potassium citrate, Allopurinol) — Eligible patients, who fulfilled the study criteria, will be instructed For; Oral alkalinization therapy
  * Potassium citrate 20 mEq three times daily
  * Hyperuricosuric patients (24-hours urine uric acid more than 750 mg/day in male and more than 650mg/day in females) will receive:
  Allopurinol, a competitive inhibitor of xanthine oxidase, in a dose of 300 mg daily.
  Other Names: systemic chemolysis
Behavioral: Life style modification — Eligible patients, who fulfilled the study criteria, will be also instructed for;
  Adequate fluid intake in order to maintain urine volume between 2-3 L per day.
Dietary Supplement: Dietary recommendations (decrease purine rich diet as red meat and fish, increase vegetables) — Eligible patients, who fulfilled the study criteria and they are hyperuricosuric (24-hours urine uric acid more than 750 mg/day in male and more than 650mg/day in females) will be also instructed for; Dietary modification will be advised in the form of decrease purine rich diet as red meat and fish, increase vegetables.

SUMMARY:
The aim of the study is to evaluate the predictors of success of oral dissolution therapy in radiolucent renal stones in a large series of patients from a tertiary referral center in order to define the optimum case scenarios where oral dissolution therapy could be implemented.

DETAILED DESCRIPTION:
Patients with renal stones, seen through the outpatient clinic in the urology department or post primary intervention for renal stones, will be assessed to see if the patient satisfies all inclusion and exclusion criteria. Patients who are meeting these criteria will be asked to participate in this prospective study. If they agree, they will be asked to sign an informed consent.

Baseline patients' assessment will include;

* Full history taking including

  * Previous stone history regarding presentation and management
  * Previous trial oral dissolution therapy for renal stones and their compliance to the treatment
  * Previous GIT surgery
  * History of chronic medical or metabolic illness e.g; DM
* Clinical examination including

  o Body mass index (BMI)
* Laboratory investigations including;

  * Urine analysis (urine PH)
  * 24 hours urine testing for uric acid and citrate
  * Urine culture
  * Serum creatinine
  * Random blood sugar (RBS)
  * Serum uric acid
  * Serum calcium, phosphorus and magnesium.
* Initial radiological evaluation will include

  * Renal ultrasonography (US)
  * Plain X-rays to exclude the presence of calcification in the targeted stone.
  * Non Contrast Computed Tomography (NCCT) on the abdomen and pelvis.
  * MAG3 diuretic renogram

(All NCCT studies will be performed with multislice helical CT scanners, NCCT images will be obtained from above the kidneys through the bladder base. For each renal stone, its location will be recorded, its size will be measured using the largest dimension from length (L), width (W) and height (H) on axial and coronal reformat images. Its mean density will be recorded by measurement using region of interest just smaller than the stone. Associated hydronephrosis proximal to the stone will be also evaluated (Nakada et al 2000).)

Patient will receive the allocated instructions and medications

Patients' follow up (The aim at follow up is to monitor the urinary PH with adjustment of the dose of potassium citrate and also to assess the compliance of the patients regarding the dietary recommendations and the medications)

* After 2 weeks, 4 weeks, 8 weeks and 12 weeks.

  - the most important parameter will be assessed is the urinary PH every two weeks. The target urinary PH should be kept between6.5 to 7.0, the dose of potassium citrate should be adjusted to achieve this value.
* Patients' compliance to medications intake and the instruction of fluid intake and dietary modification.

ELIGIBILITY:
Inclusion Criteria:

* Patients' criteria:

  1. Ability to give informed consent.
  2. Age more than 18 years.
  3. Absence of significant hydronephrosis, serious urinary tract infection, congenital anomalies or distal ureteric obstruction in the affected renal unit.
  4. Normal cardiac, hematological, and renal functions.
* Stone criteria:

  1. Primary or recurrent renal stone.
  2. Patients with residual renal stones after primary intervention whether open surgery, endoscopic or ESWL.
  3. Peripheral calyceal stones or stone in the renal pelvis with no significant hydronephrosis.
  4. Stone size less than 3 cm in maximum diameter
  5. Stones with radiodensity less than 600 Hounsefield units attenuation in Non Contrast Computed Tomography (NCCT).

Exclusion Criteria:

* Patients' criteria:

  1. Inability to give informed consent.
  2. Age less than 18 years
  3. Patients with unremitting pain or serious urinary tract infection.
  4. Presence of significant hydronephrosis, congenital anomalies or distal ureteric obstruction in the affected renal unit.
  5. Abnormal cardiac, hematological or renal functions.
* Stone criteria:

  1. Obstructing stone in the renal pelvis with significant hydronephrosis.
  2. Assumption of presence of calcium stones by presence of calcification in the stone in plain X-rays.

     -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be change in stone surface area after 3 months of the determined protocol | participants will be followed for the duration of medical treatment which is specified to be 3 months
  The stone surface area will be measured using the formula; Surface area = length X width X 0.25 X (22/7) Comparison of the stone surface area in relation to the initial surface area will be done.

SECONDARY OUTCOMES:
Assessment of the predictors of response (more than 50% reduction in the surface area of the stone) to medical treatment | participants will be followed for the duration of medical treatment which is specified to be 3 months
  The percent reduction of stone surface area will be calculated using the formula:
  Surface area = length X width X 0.25 X (22/7)
  Categorization of the patients into three groups will be done:
  * Patients who achieved 50% or more reduction in the stone surface area will be considered responsive and would be counseled for another 3 months therapy.
  * Patients with partial response, less than 50% reduction in stone surface area will be counseled for auxiliary procedure based on stone criteria e.g. ESWL.
  * Patients with no response/ serious renal infections or serious treatment adverse effects will be considered for other interventional treatment modalities.
  In the responders groups, factors predicting the success of treatment will be determined

OTHER OUTCOMES:
The cost efficiency of this procedure | participants will be followed for the duration of medical treatment which is specified to be 3 months
  Cumulative cost of medical treatment, including cost of medications and cost savings of sparred medical resources of interventional treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Shokeir, MD, Study Chair — Urology And Nephrology Center, Mansoura University, Mansoura
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt